CLINICAL TRIAL: NCT04050930
Title: Mastication Involvement in Postprandial Thermogenesis Via Autonomic Nervous System Activation in Normal Weight and Obese People
Brief Title: Mastication and Energy Expenditure in Normal Weight and Obese People
Acronym: MASTICAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Centre de Recherche en Odontologie Clinique (CROC), Faculté Dentaire (Unknown); CHU Saint Etienne Nord, Service de Physiologie Clinique et Exercice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHRC IR 2010 BOIRIE; 2018-A00724-51 (Other: ANSM)
Record Dates: First submitted 2019-07-26; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Nutrition; Mastication
Keywords: mastication; postprandial thermogenesis; autonomic nervous system; cephalic phase reflex; food texture
MeSH Terms: interventions — Mastication

STUDY DESIGN:
Intervention Model Description: each volunteer will participate to the whole protocol, that is 5 recording sessions, which, except the first session, will be organized in a random order for each volunteer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight, normo-dented (Experimental): healthy young male presenting a good oral health ad a normal weight
  Interventions: Other: Mastication
- Obese, normo-dented (Experimental): healthy young male presenting a first level of obesity, and a good oral health
  Interventions: Other: Mastication

INTERVENTIONS:
Other: Mastication — Simultaneous recordings of postprandial thermogenesis (gas exchange), cardiac activity (ECG), masticatory muscle contraction (EMG), and blood collection, during alternating periods of no-mastication or mastication of natural foods or chewing gums of different hardness

SUMMARY:
The objective of the study is to analyze the specific role of physical properties of food and mastication in the cephalic phase reflex of thermogenesis, and the involvement of the autonomic nervous system in the implementation of this reflex.

The hypothesis of the study is that oral stimulation elicited by food properties during mastication can generate changes in the amplitude of variation of thermogenesis, and that these changes are distinct from those attributable to the thermal effect of food during digestion.

DETAILED DESCRIPTION:
A group of 12 subjects presenting a normal weight and a group of 12 obese subjects, with a good general health and a good dental state will be constituted. They will participate to 5 different recording sessions during which they will be invited to chew and spit out foods and chewing gums of different hardness. During recording sessions with mastication and no-mastication periods, gas exchange (O2 concentration), cardiac activity (electrocardiography) and muscular activity of masticatory muscles (electromyography) will be recorded. Blood samples will be collected during one of the sessions to analyse the kinetic of appearance of some hormones in the blood compartment during or just after mastication. The selected hormones are involved in the eating behaviour and its regulation (ghrelin, peptide C, peptide YY and glucose-like peptide 1). From these recordings, energy expenditure, heart rate variability, intensity of masticatory muscle contraction, and hormone blood appearance will be analysed in link with the nature and hardness of the food chewed. Since the food bolus is spit out after mastication (without any swallowing = sham-feeding), the changes observed in theses variables will be directly attributed to sensory information coming from oral cavity during mastication. Food choice and sport activity of each volunteer will be taken into account to compare the results obtained for the two groups (normal weight and obese).

The work will produce more data and evidence on the contribution of oral signals attributable to the food in the regulation of the energy balance. The results will also bring more knowledge on the involvement of the autonomic nervous system. Comparison of the results obtained for the two groups (normal weight and obese people), will bring some positive outcomes which could be useful in the fight against obesity.

ELIGIBILITY:
Inclusion criteria :

19 < body mass index < 25 kg/m2 for the normal weight group 30 < body mass index < 35 kg/m2 for the obese group Good general health

Exclusion criteria :

* sport activity
* Smoking in the 6 months before the beginning of the study
* Regular alcohol consumption (more than 4 unit/day)
* Medication that may interfere with the results of the study (beta-blockers, corticoids, anti-inflammatories, thyroid hormone, insulin, antiarrhythmics) or that may have an effect on salivation or muscular activity
* Oral or dental pathology (including pain), current oral care
* Orthodontic treatment in the 3 years before the study
* Weigh gain or weight loss of more than 10% in the 3 last months
* Thyroid disturbance
* High blood pressure
* Cardiac activity anomaly
* Anomaly for one of the biological elements : complete blood count, fasting blood glucose, glycated haemoglobin, thyroid hormone (TSH), sedimentation rate > 8mm, CRP rate > 10ml/L
* Allergies, intolerance or disgust for one of the food tested

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measure of energy expenditure by Indirect calorimetry | 1 hour 30 minutes
  effect of mastication without swallowing on energy expenditure (kcal/24h) in normal weight and obese people. This will be measured by indirect calorimetry (Under Canopy of the system Fitmate)
Measure of cardiac activity | 1 hour 30 minutes
  effect of mastication without swallowing on cardiac activity (R-R interval) in normal weight and obese people measured by electrocardiogram
Measure of masticatory muscle activity | 1 hour 30 minutes
  effect of mastication without swallowing on masticatory muscle activity (microvolt.s in normal weight and obese people measured by electromyography
Estimate of the hormonal response | 1 hour 30 minutes
  effect of mastication without swallowing on hormonal response in normal weight and obese people. This will be estimate by their concentration and their kinetic of appearance in the blood compartment, and by comparisons of concentration values with basal level, also expressed in "area under the curve" values.

SECONDARY OUTCOMES:
effect of sensory information from oral cavity on energy expenditure by Indirect calorimetry | 1 hour 30 minutes
  effect of various oral information coming from oral cavity during mastication (food hardness, type of food…) on energy expenditure (kcal/24h) in normal weight and obese people. This will be measured by indirect calorimetry (Under Canopy of the system Fitmate)
effect of sensory information from oral cavity on cardiac activity | 1 hour 30 minutes
  effect of various oral information coming from oral cavity during mastication (food hardness, type of food…) on cardiac activity (R-R interval) in normal weight and obese people. This will be measured by electrocardiogram.
effect of sensory information from oral cavity on hormonal response | 1 hour 30 minutes
  effect of various oral information coming from oral cavity during mastication (food hardness, type of food…) on hormonal response in normal weight and obese people. This will be estimate by their concentration and their kinetic of appearance in the blood compartment, and by comparisons of concentration values with basal level, also expressed in "area under the curve" values.
effect of sensory information from oral cavity on masticatory muscle activity | 1 hour 30 minutes
  effect of various oral information coming from oral cavity during mastication (food hardness, type of food…) on masticatory muscle activity (microvolt.s) in normal weight and obese people. This will be measured by electromyography
cardiac activity while sleeping measured by electrocardiogram | 8-10 hours (night)
  evaluation of the general tonus of the autonomic nervous system in normal weight and obese people (R-R interval measured by electrocardiogram)
cardiac activity (frequency analysis) while sleeping measured by electrocardiogram | 8-10 hours (night)
  evaluation of the general tonus of the autonomic nervous system in normal weight and obese people
global characterization of sport activity | 4 consecutive days
  evaluation of the mean energy expenditure in link with physical activity (kcal/time unit) to have a global characterization of the volunteer. This will be done by the app WellBeNet wich contains eMouv for sport activities.
global characterization of food choices | 4 consecutive days
  evaluation of the mean energy expenditure in link with food choices and food habits (food portion, score), to have a global characterization of the volunteer. This will be done by the app WellBeNet wich contains NutriQuantic for food choices

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Professor, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France